CLINICAL TRIAL: NCT05513118
Title: Evaluation of the Relationship Between Menopause and Periodontal Health With Biochemical and Microbiological Parameters
Brief Title: Menopause and Oral Health
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gülnur Emingil, Prof. Dr., Ege University
Other Study IDs: TOA-2020-21085
Record Dates: First submitted 2022-08-21; First posted 2022-08-24 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Menopause; Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-menopausal women
  Interventions: Diagnostic Test: Periodontal clinical examination and gingival crevicular fluid, saliva, dental plaque, serum sampling
- Regularly mensturating women
  Interventions: Diagnostic Test: Periodontal clinical examination and gingival crevicular fluid, saliva, dental plaque, serum sampling

INTERVENTIONS:
Diagnostic Test: Periodontal clinical examination and gingival crevicular fluid, saliva, dental plaque, serum sampling — Probing pocket depth was defined as the distance in millimeters from the gingival margin to the base of the gingival sulcus measured using a manual probe (Michigan 0 probe with Williams Markings) in all the teeth present except for third molars. Similarly, clinical attachment level (CAL) was measured as distance from cementoenamel junction to the base of pocket and recorded manually to the nearest millimeter marking on probe.
  1 mililiter of saliva was obtained by each participant. Subgingival dental plaque was collected with sterile endodontic paperpoints from mesial sides of each natural teeth without a prostethic restoration. Gingival crevicular fluid samples were collected with absorbent paper strips. Serum samples were also collected at the time of visit.

SUMMARY:
Menopause is characterized by major physiological and concomitant psychological changes. The study aimed to evaluate the association between oral health parameters, bone mineral density (BMD) and physiological or psychological symptoms in post-menopausal women (PMW), compared with regularly menstruating women (RMW). Inflammatory biomarker levels in gingival crevicular fluid, saliva, serum and determination of microbial niches in subgingival plaque samples were further aimed. The participants were asked to complete the Women's Health Questionnaire to measure emotional and physical well-being.

A total of 148 women (PMW, n=76,RMW, n=72) received a comprehensive medical assessment and a full-mouth oral examination. The corresponding bone mineral density (BMD) and body mass indices (BMI) were obtained from their medical records.

ELIGIBILITY:
Inclusion Criteria:

* Being 35-65 years of age
* Having history of spontaneous amenorrhea for the last 12 months for PMW.
* Lack of irregularity in menstrual cycles during the past 12 months for RMPW.
* Possessing at least 10 natural teeth without any prosthetic restoration

Exclusion Criteria:

* History of antibiotics use in last 3 months
* Ongoing cancer therapy
* Presence of oral ulcers or acute infectious disease
* Presence of diabetes mellitus

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population comprised of two main groups as postmenopausal women (PMW) and regularly menstruating women (RMW). The women in the PMW group were included if they were under 65 years of age and had a history of spontaneous amenorrhea for the last 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Periodontitis | 1 month
  Interdental attachment loss is detectable at ≥2 non-adjacent teeth, or buccal/oral attachment loss ≥3 mm with pocketing >3 mm at ≥2 adjacent teeth were present.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Dentistry, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided